CLINICAL TRIAL: NCT03980418
Title: Comparative Study of DaTSCAN ™ Cerebral SPECT Recorded by Conventional Anger Cameras and Semiconductor Camera (VERITON-CT ™)
Brief Title: Evaluation of a Semiconductor Camera for the DaTSCAN™ Exam
Acronym: VERIDAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, MD, PhD, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PSS2019/VERIDAT-VERGER-VS
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; DaTSCAN™ SPECT/CT scintigraphy; Semiconductor CZT camera "with large field"
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all included patients will have the same procedure (Experimental): After the conventional DaTSCAN SPECT/CT exam in conventional camera, all patients included will have two recordings of DaTSCAN SPECT/CT in semiconductor CZT (cadmium zinc telluride) camera; one focused on the striatum and the other focused on the total brain
  Interventions: Procedure: DaTSCAN SPECT/CT in VERITON-CT camera

INTERVENTIONS:
Procedure: DaTSCAN SPECT/CT in VERITON-CT camera — the intervention is based on two recordings in camera VERITON-CT ; the first, in focus striatum mode and the second in brain focus mode

SUMMARY:
The semiconductor (cadmium-zinc-telluride, CZT) cameras significantly increase detection sensitivity in Single Photon Emission Computer Tomoscintigraphy (SPECT)(1) . The clinical routine applications of these cameras are today mainly limited to myocardial tomoscintigraphy with CZT dedicated cameras. Several studies whose one was done in Hospital of Nancy, made it possible to demonstrate a good diagnosis agreement between conventional cameras and semiconductor cameras in this indication, with better image quality obtained with semiconductor cameras (2). Today, so-called "wide field" semiconductor cameras are available in the clinic and allow for any type of SPECT examination. A comparative study between conventional and semiconductor cameras has been conducted for bone scintigraphy, and shows diagnostic superiority with this new type of camera (3).

In addition, the new VERITON-CT ™ (Spectrum Dynamics Medical) camera has 12 mobile CZT-based detectors positioned around the patient allowing tomographic acquisitions and focusing the acquisition on the organ studied. This camera has a sensitivity of detection higher than that of conventional cameras and thus reduces the activity injected into the patient and / or the recording time.

To date, no study has compared the two types of cameras in nuclear neurology and in particular, for the SPECT DaTSCAN ™ imaging of the pre-synaptic dopaminergic pathway.

DaTSCAN ™ exam is used in clinical routine:

1. for the diagnosis of Parkinson's disease or related diseases when in doubt with an essential tremor (4) or
2. if suspicion of Lewy body disease, if in doubt with Alzheimer's disease (5). If the interpretation of DaTSCAN ™ exam is first visual, the quantification may increase accuracy diagnosis (6). Also, the database creation specific to each type of camera is recommended(7).

The purpose of this study is to compare the diagnostically relevant informations and the quantitative analysis provided by the DaTSCAN™ SPECT, recorded on the conventional camera and recorded on the semiconductor camera VERITON-CT™

DETAILED DESCRIPTION:
The clinical study is monocentric, interventional, non randomized, with minimal risk and constraints.

All patients going to the nuclear medicine department for a DaTSCAN exam will be able to participate in this study if they understood study informations given by the physician and if they signed the inform consent.

In first, patients will have a DaTSCAN™ SPECT on a conventional camera and after, they will have DaTSCAN™ SPECT on VERITON-CT™ camera with two records: one in focus striatum mode and the second in focus brain mode.

The attenuation correction will be made with the computer tomography (CT) recorded at the same time as the SPECT (SPECT/CT)

ELIGIBILITY:
Inclusion Criteria:

* all patients over 18 years sent to Datscan SPECT/CT
* patients understanding and having signed the informed consent form.
* without contraindication to have the scintigraphy
* patient subject to a medical benefits scheme

Exclusion Criteria:

* known allergy to the one of the components of Datscan
* pregnant, parturient or breastfeeding woman
* major person under legal protection (any form of public guardianship)
* major person unable to express consent
* person deprived of liberty due to judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Degree of concordance (Kappa) of the exams results of different records | 16 months
  comparison between the exam results (positive diagnosis of Parkinson disease or Lewy bodies dementia versus differential diagnosis) in conventional camera and the one obtained with the VERITON-CT in striatum focus mode

SECONDARY OUTCOMES:
Degree of concordance (Kappa) of the exams results of different recordings | 16 months
  comparison between the exam results (positive diagnosis of Parkinson disease or Lewy bodies dementia versus differential diagnosis) in conventional camera and the one obtained with the VERITON-CT in brain focus mode

OTHER OUTCOMES:
Degree of concordance (Kappa) of the exams results of different recordings | 16 months
  comparison between the exam results (positive diagnosis of Parkinson disease versus differential diagnosis) in conventional camera and the one obtained with the VERITON-CT in striatum focus mode
Degree of concordance (Kappa) of the exams results of different recordings | 16 months after the first enrollment
  comparison between the exam results (positive diagnosis of Lewy bodies dementia versus differential diagnosis) in conventional camera and the one obtained with the VERITON-CT in striatum focus mode
ratios of uptake obtained with conventional camera and on the striatum focus record with VERITON-CT | immediately after SPECT-CT exam
  the uptake ratios are:caudate nuclei/occipital cortex, putamen/occipital cortex, to the right and caudate nuclei/medium cingulate cortex, putamen/medium cingulate cortex to left, obtained with conventional camera and on the striatum focus record with VERITON-CT camera
quality scores of images from conventional camera and from VERITON (striatum) | immediately after SPECT-CT exam
  0= very bad quality and impossible to do a diagnosis, 1=bad quality and difficult diagnosis, 2= medium quality, 3 = good quality and 4= excellent quality
recording activity in striatal area for the images from conventional camera and from VERITON (striatum) | immediately after SPECT-CT exams
  recorded activities will be reported by injected MBq for the images obtained with the conventional camera and with VERITON striatum focus record
score of diagnosis agreement for the images interpretation by 3 physicians | 18 months
  The agreement will be between conventional record and striatum focus record with VERITON camera
uptake ratios on the conventional record and on the focus brain record with VERITON | after each SPECT/CT exams
  the uptake ratios are:caudate nuclei/occipital cortex, putamen/occipital cortex, to the right and caudate nuclei/medium cingulate cortex, putamen/medium cingulate cortex to left, obtained with conventional camera and on the brain focus record with VERITON-CT camera
quality scores of images from conventional camera and from VERITON (brain) | immediately after SPECT-CT exams
  0= very bad quality and impossible to do a diagnosis, 1=bad quality and difficult diagnosis, 2= medium quality, 3 = good quality and 4= excellent quality
recording activity in striatal area for the images from conventional camera and from VERITON (brain) | 18 months
  recorded activities will be reported by injected MegaBecquerel (MBq) for the images obtained with the conventional camera and with VERITON brain focus record
diagnosis agreement for the interpretation by 3 physicians between conventional and VERITON (brain) | 18 months
  The agreement will be between conventional record and brain focus record with VERITON camera

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU of Nancy, Vandœuvre-lès-Nancy, France